CLINICAL TRIAL: NCT06742658
Title: A Retrospective Study on the Safety of the Rapid Move Following Outpatient Surgery and the Characteristics of Patients in the Rapid Move
Brief Title: Rapid Move Following Outpatient Surgery: Safety and Patient Characteristics
Acronym: OUTSIDE
Status: Not yet recruiting | Type: Observational
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Collaborators: University Ghent (Other)
Responsible Party: Principal Investigator, Ella Hemie, studiecoordinator, PhD student, Algemeen Ziekenhuis Maria Middelares
Other Study IDs: MMS.2024.079
Record Dates: First submitted 2024-12-13; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Recovery
Keywords: Postoperative recovery; PACU; Rapid Move

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients undergoing an outpatient procedure eligible for the Rapid Move.: Patients who went to the Rapid Move after their outpatient procedure. Eligible procedures are: gastroscopy, coloscopy, vasectomy, scrotal surgery, circumcision or other minor penile surgery, intravesical Botox, insertion or removal of eardrum tubes in adults, sinus irrigation in adults, sleep endoscopy, bronchoscopy, removal of osteosynthetic material in the lower leg and foot, and tooth extraction (including wisdom teeth) and upper-forearm orthopaedic surgery (excluding prosthetic surgery).
  Interventions: Other: Rapid Move

INTERVENTIONS:
Other: Rapid Move — A short-stay PACU where patients recover from anaesthesia, are continuously monitored, and prepared for discharge within an hour after surgery.

SUMMARY:
A descriptive, retrospective cohort study will be conducted to gain insight in the safety of the Rapid Move. The trial will include a group of Rapid Move patients, who were transferred to the Rapid Move after their outpatient surgery and subsequently discharged home. The Rapid Move is a short-stay PACU where patients recover from anaesthesia, are continuously monitored, and prepared for discharge within an hour after surgery.

DETAILED DESCRIPTION:
The Rapid Move, a short-stay PACU unit, was implemented at General Hospital Maria Middelares in Ghent, Belgium. The Rapid Move is designed to alleviate the bottleneck in the day surgery unit. Overcrowding in the PACU, caused by limited space in the day surgery unit, resulted in delays in patient discharge despite patients meeting discharge criteria. The Rapid Move is designed for brief, intensive follow-up care, similar to the PACU, with continuous monitoring and a nurse-to-patient ratio of 2:9. An analysis of the occupancy rate of the PACU and the Rapid Move indicates that, despite overcrowding in the PACU, the Rapid Move is still underutilised. Despite the extensive research on PACU bypassing, to our knowledge, no research has been conducted on the safety of the Rapid Move, a short-stay PACU where patients recover from anaesthesia, are continuously monitored and prepared for discharge within an hour after surgery. The aim of this retrospective cohort study is to gain insight in the safety of the Rapid Move as an alternative postoperative pathway for outpatients.

Furthermore, the underutilisation of the Rapid Move, despite the overcrowding of the PACU, has highlighted the need to develop a patient profile of eligible patients for the Rapid Move, with the intention to expand the selection criteria for the Rapid Move and optimise its capacity.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15 years or older;
* Patients who went to the Rapid Move after their outpatient procedure. Eligible procedures are: gastroscopy, coloscopy, vasectomy, scrotal surgery, circumcision or other minor penile surgery, intravesical Botox, insertion or removal of eardrum tubes in adults, sinus irrigation in adults, sleep endoscopy, bronchoscopy, removal of osteosynthetic material in the lower leg and foot, and tooth extraction (including wisdom teeth) and upper-forearm orthopedic surgery (excluding prosthetic surgery).

Exclusion Criteria:

* Inpatients defined as a patient who is formally admitted (or "hospitalized") to an institution for treatment and/or care and stays for a minimum of one night in the hospital or other institution providing inpatient care;
* Patients undergoing emergency procedures.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include an intervention group with all consecutive patients, aged 15 years or older, who went to the Rapid Move after their outpatient procedure between 1 December 2023 and 1 December 2024 in general hospital Maria Middelares, Ghent, Belgium (Rapid Move patients).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
30-day readmission | Up to 30 days after hospital discharge.
  The 30-day readmission rate is defined as the number of patients with an unplanned emergency hospital readmission, including emergency department (ED) visits with or without hospital readmission, occurring between the time the patient is discharged from the hospital after their outpatient surgery (index hospital admission) and 30 days after the surgery. An admission to a non-acute care facility is not considered a readmission. A readmission must be clinically related to the index hospital admission. The term 'clinically related' is defined as meaning that the underlying reason for readmission is plausibly related to the care rendered during or immediately following a prior hospital admission. A clinically related readmission may have resulted from the process of care and treatment during the prior admission or from a lack of post-admission follow-up, rather than from events that occurred after the prior admission within a specified readmission time interval that are unrelated to the p

SECONDARY OUTCOMES:
Complications | Up to 30 days after hospital discharge.
  Readmission reason, classified using the International Classification for Diseases (ICD)-11.
Length of Stay | Minutes, up to 4 hours.
  The time between the arrival at the Rapid Move unit and the time of hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ella Hermie, MSc, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No